CLINICAL TRIAL: NCT00736892
Title: Acute Lung Injury: Epidemiology and Natural History. The ALIEN Study
Brief Title: Incidence of Acute Lung Injury: The Alien Study
Acronym: ALIEN
Status: Completed | Type: Observational
Sponsor: Villar, Jesus, M.D. (Individual)
Responsible Party: Principal Investigator, Jesus Villar, Director of Research, Dr. Negrin University Hospital
Other Study IDs: 2008-0915-EPI
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Acute Lung Injury
Keywords: Acute lung injury; Acute respiratory distress syndrome; Mechanical ventilation; Prognosis; Definitions
MeSH Terms: conditions — Acute Lung Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A: All patients meeting the American European Consensus definition of acute lung injury will be included, regardless of etiology of respiratory failure. Specifically, all patients with rapid onset of acute lung injury not of cardiac origin (no indication of heart failure or a pulmonary capillary wedge pressure of greater than 18 mmHg, with pulmonary infiltrates in all four quadrants and a PaO2/FIO2 of > 200 to <300 mmHg or ≤ 200 mmHg.

SUMMARY:
Acute lung injury is a clinical syndrome of rapid onset of acute respiratory failure. It represents a significant public health issue. Patients with acute lung injury require admission into critical care units for advanced life support and utilize considerable health care resources. Published epidemiological studies on acute lung injury in the last 20 years are difficult to compare because they used different definitions and length of time for evaluation. Less than five studies have collected information for an entire year, and none of them have evaluated the degree of oxygenation failure under standard settings. We will perform a one-year prospective audit of all patients admitted with acute lung injury in almost 40 ICUs in Spain.

DETAILED DESCRIPTION:
Acute lung injury (ALI) is a clinical syndrome of rapid onset of non-cardiogenic pulmonary edema manifested clinically by hypoxemia (PaO2/FiO2≤300 mmHg) and bilateral pulmonary infiltrates. When the hypoxemia is severe (PaO2/FiO2≤200 mmHg) it is termed the acute respiratory distress syndrome (ARDS). It represents a significant public health issue. Patients with ALI or ARDS require admission into critical care units for advanced life support and utilize considerable health care resources.

An immense plethora of translational knowledge has been acquired since the first description of ARDS in 1967. However, estimates of the incidence of ARDS and ALI have varied widely, and the true magnitude of this health problem still remains unclear. Current estimates of the incidence of ALI/ARDS range from 15 to 80 cases per 100.000 population, or almost 40.000 cases per year in Spain. Combined mortality rates for ALI/ARDS range between 30-45%. ALI and ARDS occur as a complication or as the primary cause of critical illness in patients, usually after severe infection or trauma.

Published epidemiological studies on ALI and ARDS in the last 20 years are difficult to compare. Some reports have used different definitions for ALI and ARDS and others have evaluated the incidence during a short period of time (from days to several weeks) and then extrapolated their data to estimates of a one-year incidence. Very few studies have collected information for an entire year, and none of them have evaluated the degree of hypoxemia under standard ventilatory settings, as it has been proposed recently by the HELP Network (Am J Respir Crit Care Med 2007; 176:795-804).

As a result, we propose to perform a one-year prospective audit of all ALI and ARDS patients managed in 40 ICUs from 17 Spanish provinces (15 provinces in the mainland and 2 provinces in the Canary Islands). We intend to collect data from all patients admitted with or developing ALI/ARDS with the aim to understand the epidemiology and natural history of acute lung injury. These provinces are scattered through the Spain and are representative of the demographic differences across the country.

ELIGIBILITY:
Inclusion Criteria:American-European Consensus Conference Definition criteria for acute lung injury:(i) rapid onset of acute lung injury not of cardiac origin; (ii) bilateral pulmonary infiltrates on chest X ray; (iii) PaO2/FIO2<300 mmHg.

Exclusion Criteria: None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted into intensive care units of participating hospitals across Spain meeting the American-European Consensus Conference definition of acute lung injury.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2010-03 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Incidence of acute lung injury and the acute respiratory distress syndrome | 12 months

SECONDARY OUTCOMES:
Risk factor associated with acute lung injury | 12 months
Mortality rates of acute lung injury, acute respiratory distress syndrome and combined | 12 months
Identification of clinical data associated with the highest or lowest mortality | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jesus Villar, MD, PhD, Principal Investigator — Hospital Universitario Dr. Negrin, Las Palmas, Spain; Robert M Kacmarek, PhD, Principal Investigator — Massachusetts General Hospital, Boston, USA
Locations (1):
- Hospital Universitario Dr. Negrin, Las Palmas de Gran Canaria, Canary Islands, Spain

REFERENCES:
- [Derived] Villar J, Gonzalez-Martin JM, Ambros A, Mosteiro F, Martinez D, Fernandez L, Soler JA, Parra L, Solano R, Soro M, Del Campo R, Gonzalez-Luengo RI, Civantos B, Montiel R, Pita-Garcia L, Vidal A, Anon JM, Ferrando C, Diaz-Dominguez FJ, Mora-Ordonez JM, Fernandez MM, Fernandez C, Fernandez RL, Rodriguez-Suarez P, Steyerberg EW, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. Stratification for Identification of Prognostic Categories In the Acute RESpiratory Distress Syndrome (SPIRES) Score. Crit Care Med. 2021 Oct 1;49(10):e920-e930. doi: 10.1097/CCM.0000000000005142. PMID 34259448
- [Derived] Villar J, Ambros A, Mosteiro F, Martinez D, Fernandez L, Ferrando C, Carriedo D, Soler JA, Parrilla D, Hernandez M, Andaluz-Ojeda D, Anon JM, Vidal A, Gonzalez-Higueras E, Martin-Rodriguez C, Diaz-Lamas AM, Blanco J, Belda J, Diaz-Dominguez FJ, Rico-Feijoo J, Martin-Delgado C, Romera MA, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification and Therapies of ARDS (SIESTA) Network. A Prognostic Enrichment Strategy for Selection of Patients With Acute Respiratory Distress Syndrome in Clinical Trials. Crit Care Med. 2019 Mar;47(3):377-385. doi: 10.1097/CCM.0000000000003624. PMID 30624279
- [Derived] Villar J, Martinez D, Mosteiro F, Ambros A, Anon JM, Ferrando C, Soler JA, Montiel R, Vidal A, Conesa-Cayuela LA, Blanco J, Arrojo R, Solano R, Capilla L, Del Campo R, Civantos B, Fernandez MM, Aldecoa C, Parra L, Gutierrez A, Martinez-Jimenez C, Gonzalez-Martin JM, Fernandez RL, Kacmarek RM; Stratification and Outcome of Acute Respiratory Distress Syndrome (STANDARDS) Network. Is Overall Mortality the Right Composite Endpoint in Clinical Trials of Acute Respiratory Distress Syndrome? Crit Care Med. 2018 Jun;46(6):892-899. doi: 10.1097/CCM.0000000000003022. PMID 29420341
- [Derived] Villar J, Blanco J, del Campo R, Andaluz-Ojeda D, Diaz-Dominguez FJ, Muriel A, Corcoles V, Suarez-Sipmann F, Tarancon C, Gonzalez-Higueras E, Lopez J, Blanch L, Perez-Mendez L, Fernandez RL, Kacmarek RM; Spanish Initiative for Epidemiology, Stratification & Therapies for ARDS (SIESTA) Network. Assessment of PaO(2)/FiO(2) for stratification of patients with moderate and severe acute respiratory distress syndrome. BMJ Open. 2015 Mar 27;5(3):e006812. doi: 10.1136/bmjopen-2014-006812. PMID 25818272